CLINICAL TRIAL: NCT06347809
Title: DNA Methylation in Adenocarcinoma of the Prostate: Analysis of Validated Biomarkers in Urine
Status: Terminated | Type: Observational
Why Stopped: Closed to consolidate enrollment under another related study
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-006343; NCI-2024-01225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-006343 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-03-15; First posted 2024-04-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prostate Adenocarcinoma; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Participants can choose whether they permit their urine samples to be stored and used in future cancer research at Mayo Clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: PHASE I: Participants undergo urine sample collection on study.
  PHASE II: Participants undergo standard prostate massage and collection of prostatic fluid and urine samples on study.
  All participants complete a questionnaire and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study explores the potential use of DNA markers in the detection of prostate cancer and patient perceptions of this screening approach and other current or future prostate cancer screening and diagnostic tests.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the accuracy of MDM candidates (individually and in combination) assayed from urine and prostatic fluid (collected following digital prostate massage) for detection of CAP.

OUTLINE: This is an observational study.

PHASE I: Participants undergo urine sample collection on study.

PHASE II: Participants undergo standard prostate massage and collection of prostatic fluid and urine samples on study.

All participants complete a questionnaire and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * Patient is 18 years or older

  * Patient has a histologically confirmed diagnosis of prostatic carcinoma/adenocarcinoma with a corresponding Gleason score OR is scheduled for a prostate biopsy for an elevated Prostate Specific Antigen (PSA), palpable prostate nodule, an abnormal imaging finding, or worrisome PSA velocity

Exclusion Criteria:

* * Patient has had a transplant prior to sample collection

  * Patient has had Androgen (e.g. Flutamide, Androcur, Casodex, Nilandron) or Luteinizing hormone-releasing hormone (LHRH) (e.g. Lupron, Zoladex) therapy
  * Patient has transurethral instrumentation (cystoscopy, placement of urinary catheter) within the 7 days prior to sample collection
  * Patient has chronic indwelling urinary catheter
  * Patient has had a urinary tract infection within the 14 days prior to sample collection
  * Patient has immunotherapy (e.g. Kwon study drugs) for prostate cancer prior to sample collection
  * Patient has a history of bladder cancer
  * Patient has had a biopsy within the last 6 weeks (excluding non-melanoma skin biopsies) of sample collection
  * Patient has had surgery to completely remove current target pathology prior to sample collection
  * Patient has a prior history of prostate carcinoma/adenocarcinoma
  * Patient has received chemotherapy class drugs (e.g. Docetaxel, Methotrexate) within the 5 years prior to sample collection
  * Patient has received therapeutic radiation prior to sample collection
  * Patient has had focal ablation [e.g. High-intensity focused ultrasound (HIFU) or cryoablation] of prostate cancer prior to sample collection
  * Patient has known primary cancer outside of the prostate within the last 5 years (not including basal cell or squamous cell skin cancers) of sample collection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of prostate carcinoma/adenocarcinoma with a corresponding Gleason score OR is scheduled for a prostate biopsy for an elevated PSA, palpable prostate nodule, an abnormal imaging finding, or worrisome PSA velocity.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of methylated DNA markers (MDMs) for detection of cancer of the prostate (CAP) | Baseline
  Assessed by instances of CAP detected using MDMs assayed from urine (Phase I) and from urine and prostate fluid (collected following digital prostate massage for participants in Phase II) for detection of CAP.

SECONDARY OUTCOMES:
Accuracy of CAP detection | Baseline
  Assessed by instances of CAP detected and confirmed using MDMs assayed from urine and prostate fluid.
Comparison of sample volumes | Baseline
  Variability of sample volumes will be assessed for DNA and MDM yield.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Kisiel, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials